CLINICAL TRIAL: NCT01372449
Title: A Multi-site Double-blind Placebo-controlled Trial of Memantine Versus Placebo in Children With Autism Targeting Memory and Motor Planning
Brief Title: A Multi-site Double-blind Placebo-controlled Trial of Memantine Versus Placebo in Children With Autism (MEM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evdokia Anagnostou (Individual)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Rush University Medical Center (Other); Nationwide Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Evdokia Anagnostou, Clinician Scientist, Anagnostou, Evdokia, M.D.
Organization: Anagnostou, Evdokia, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111576
Record Dates: First submitted 2011-06-02; First posted 2011-06-14 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Psychopharmacology; Clinical Trial; Children
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (Active Comparator)
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Memantine will be initiated at 3 mg. The dose will be increased every week by 3 mg for a maximum of 12mg for subjects weighing ≥ 60kg, 9mg for subjects weighing ≥ 40 kg but <60 kg, and 6 mg for subjects weighing ≥ 20 kg but < 40kg.
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will attempt to study the effect of memantine, on memory, and motor praxis/expressive language skills in children with autism.

The investigators will recruit children ages 6-12 years who are verbal and meet criteria for Autism Spectrum Disorder. The children will be assessed for memory function, expressive language output and motor skills/praxis. They will then be randomized to memantine or placebo for 6 months. The effects of this medication and its safety in this population will be studied over the 6 month period.

DETAILED DESCRIPTION:
Abnormalities in the modulation of the glutamate system have been reported by multiple investigators studying animal models, post-mortem brains, and single gene disorders that have overlapping phenotypes with autism. Abnormalities in glutamatergic function have been reported in disorders affecting a variety of behavioral and neurological domains, from mood stability, to cognitive flexibility, memory, and motor function. Numerous studies have reported a variety of memory and motor deficits in children with autism. Whereas the neurobiology of such deficits is an area of active research, there is a paucity of intervention research for such deficits in autism. This study will attempt to study the effect of an N-methyl-D-aspartate receptor (NMDA) inhibitor, memantine, on memory, and motor praxis/expressive language skills in children with autism.

Methods: Children ages 6-12 years who are verbal and meet criteria for Autism Spectrum Disorder will be recruited across 2 sites. After consent, the children will be assessed for memory function, expressive language output and motor skills/praxis. They will then be randomized 1:1 to memantine versus placebo for 6 months. The effects of this medication on the above mentioned symptoms domains as well as its safety in this population will be studied over the 6 month period.

ELIGIBILITY:
Inclusion Criteria

1. Male or female outpatients 6 to 12 years of age
2. Verbal; Module 2 or 3 on Autism Diagnostic Observation Schedule (ADOS)
3. Meet Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) for Autism Spectrum Disorder. The diagnosis will be confirmed with Autism Diagnostic Interview-Revised (ADI-R) and ADOS Module 2 or 3.
4. Parents report difficulties with motor skills
5. Have a Clinician's Global Impression-Severity (CGI-S) score ≥ 4 (moderately ill) at Screening and Baseline
6. If already receiving stable nonpharmacologic educational, behavioral, and/or dietary interventions, have continuous participation during the preceding 3 months prior to Screening and will not electively initiate new or modify ongoing interventions for the duration of the study
7. Participants can be on up to 2 concomitant psychotropic medications before entering the study, provided that they have been on a stable dose for 30 days and have no plans to adjust the dose for the duration of study
8. Have normal physical examination and laboratory test results at Screening. If abnormal, the finding(s) must be deemed clinically insignificant by the Investigators
9. Prior to the conduct of any study-specific procedures, the patient must provide assent to participate in the study (if developmentally appropriate), and the parent or legal guardian must provide written informed consent
10. The patient and the patient's parent or legal guardian must be able to speak and understand English sufficiently to understand the nature of the study and to allow for the completion of all study assessments
11. The parent or legal guardian must be capable of providing reliable information about the patient's condition, agree to oversee the administration of study drug, and accompany the patient to all clinic visits

Exclusion Criteria:

1. Patients born prior to 35 weeks gestational age
2. Patients with any primary psychiatric diagnosis other than autism at Screening: a history of Attention Deficit Hyperactivity Disorder (ADHD), bipolar disorder, psychosis, post-traumatic stress disorder, schizophrenia, or major depressive disorder
3. Patients with a medical history of neurological disease, including, but not limited to, epilepsy/seizure disorder (except simple febrile seizures), movement disorder, tuberous sclerosis, fragile X, and any other known genetic syndromes, or known abnormal MRI/structural lesion of the brain
4. Patients with a medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. Patients with evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease.
5. Patients who plan to initiate or change pharmacological or nonpharmacologic interventions during the course of the study
6. Patients on d-cycloserine or riluzole as they both target the glutamate system
7. Patients on agents that alkalinize the urine (acetazolamide, potassium citrate, and sodium bicarbonate), as they decrease the elimination of memantine
8. Patients who have received treatment with memantine in the past with no response
9. Patients with a history of hypersensitivity reaction to dextromethorphan, amantadine, or any other NMDA receptor antagonists
10. Patients unable to tolerate venipuncture procedures for blood sampling
11. Patients who, in the Investigator's opinion, might not be suitable for the study
12. Children weighing under 20 kg (to meet FDA approvals)
13. Patients with a positive pregnancy test

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2011-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Developmental Neuropsychological Assessment (NEPSY) Apraxia and Repetition of Nonsense Words Subtests | Baseline, Week 12, Week 24 (Measuring change from Baseline, middle of trial and end of trial)
  Outcome Measure is going to report a change. The NEPSY provides a developmental neuropsychological assessment for children age 3-12. It was designed to assess basic and complex aspects of cognitive capacities that are critical to children's ability to learn and be productive both in and out of school settings
Expressive Vocabulary Test (EVT) | Baseline, Week 12, Week 24 (Measuring change from Baseline, middle of trial and end of trial)

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scale - Revised | Baseline, Week 12, Week 24 (Measuring change from Baseline, middle of trial and end of trial)
  Outcome Measure is going to report a change. The Vineland Scale is a semi-structured informant interview that assesses subjects' daily functioning. It is typically administered to a caretaker/family member. This scale has been found to assess social deficits in autism and relative strengths in daily living skills.
Safety Monitoring Uniform Research Form | Screening, Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 16, Week 20, Week 24
  The SMURF consists of three parts. Part 1 contains a "General Inquiry" to obtain all information about possible physical complaints, using general probes. Part 2 comprises "Specific Inquiries" about physical complaints, organized roughly around different body systems. Part 3 concludes with a "Closing Inquiry" in which the clinician can ask about any physical or other problems he/she has pre-existing knowledge about or which he/she noticed during the rest of the inquiry.

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, M.D., Study Chair — Holland Bloorview Kids Rehabilitation Hospital; Latha V Soorya, Ph.D., Principal Investigator — Rush University Medical Center; David Grodberg, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brignell A, Marraffa C, Williams K, May T. Memantine for autism spectrum disorder. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013845. doi: 10.1002/14651858.CD013845.pub2. PMID 36006807
- [Derived] Soorya LV, Fogg L, Ocampo E, Printen M, Youngkin S, Halpern D, Kolevzon A, Lee S, Grodberg D, Anagnostou E. Neurocognitive Outcomes from Memantine: A Pilot, Double-Blind, Placebo-Controlled Trial in Children with Autism Spectrum Disorder. J Child Adolesc Psychopharmacol. 2021 Sep;31(7):475-484. doi: 10.1089/cap.2021.0010. PMID 34543081